CLINICAL TRIAL: NCT03979573
Title: Prospective Phase II Trial Evaluating Multiparametric MRI, Radiomics, MR-guided Biopsy, and Molecular Markers for Active Surveillance of Patients With Low- and Intermediate-Risk Prostate Cancer
Brief Title: Prospective Evaluation of Mp-MRI, MR-guided Biopsy, and Molecular Markers for Active Surveillance of Prostate Cancer
Acronym: PROMM-AS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5941R
Record Dates: First submitted 2018-01-28; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer
Keywords: Prospective Study; Multiparametric MRI; Radiomics; MR-guided Biopsy; Molecular Markers; Active Surveillance; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging; Radiomics

STUDY DESIGN:
Intervention Model Description: Prospective' Single-Arm, Phase-II Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Arm (Other): * PSA testing
  * Multiparametric MRI (mp-MRI)
  * Radiomics
  * MR-guided biopsy (MR-guided and systematic US-guided)
  * Molecular Markers (Histological analysis of biopsy cores)
  Interventions: Diagnostic Test: Multiparametric MRI; Diagnostic Test: Radiomics; Diagnostic Test: MR-guided Biopsy; Diagnostic Test: Molecular Markers

INTERVENTIONS:
Diagnostic Test: Multiparametric MRI — Multiparametric prostate MRI (mp-MRI)
Diagnostic Test: Radiomics — Radiomics analyses will consist of image intensity normalization, image coregistration and resampling, radiomic feature extraction, combination with clinical and molecular parameters, feature extraction and machine learning, model testing on validation and test cohorts and comparison to existing clinical risk models.
Diagnostic Test: MR-guided Biopsy — MR-guided targeted prostate biopsies as well as systematic TRUS-guided biopsies (at least 12 cores) will be performed on a fusion-guided biopsy system. The biopsy cores can either be obtained transrectal or transperineal.
Diagnostic Test: Molecular Markers — Molecular markers will be analyzed on the initial and final targeted and systematic biopsy cores. The molecular panel consists of a methylation-specific PCR and a set of highly selected markers that can be detected by immunohistochemistry. The resulting data will be prospectively recorded to enable a retrospective analysis of the prognostic value.

SUMMARY:
Active Surveillance (AS) is a treatment option in patients with favorable risk prostate cancer. According to the current guidelines patients are monitored by prostate specific antigen (PSA) testing (every 3 months) and regular re-biopsies. Due to histological reclassification and/or patient noncompliance a high number of patients discontinue AS. Nonetheless, because of an increasing number of diagnosed early stage tumors overdiagnosis and overtreatment of patients has become a major clinical problem. Therefore AS is a promising and important tool for patients with low and intermediate risk prostate cancer.

Multiparametric MRI (mp-MRI) in combination with radiomics analysis, MR-guided biopsies, and molecular markers are promising tools to optimize patient selection and observation during AS.

This prospective, single arm, multicenter phase II study evaluates mp-MRI, radiomics, MR-guided biopsies and molecular markers for AS with the primary endpoint of reducing discontinuation based on histologic reclassification.

At the end of this study the results may allow defining a MRI-based pathway to identify and monitor patients suitable for AS supported by radiomics. Thus, the high rate of discontinuation due to misclassification at initial diagnosis will be reduced.

Additionally, this strategy will allow reducing over-treatment of clinically insignificant PCA, and on the other hand, increasing early treatment of higher-risk disease. Monitoring by mp-MRI will reduce the number of prostate biopsies and cores per patient during AS, and thus increase the patient compliance. Finally, such a strategy will reduce the economic burden of treating insignificant prostate cancer.

DETAILED DESCRIPTION:
This prospective multicenter phase II study evaluates multiparametric MRI (mp-MRI), radiomics and MR-guided biopsies for Active Surveillance (AS) of men with low- and intermediate-risk prostate cancer (PCA) with the primary endpoint of reducing the rate of discontinuation of AS based on histologic reclassification in an observation period of 24 months.

Men with low- or intermediate-risk PCA diagnosed by mp-MRI followed by an MR/ultrasound fusion-guided biopsy (FUS-GB) plus systematic ultrasound-guided biopsy (SB) will be included in this study.

During the study observation period PSA values will be obtained every 3 months. After having obtained three values PSA doubling times (PSA-DT) will be calculated at every visit. In case of PSA-DT <3 years patients will get a repeat mp-MRI and in case of MRI progression a repeat targeted FUS-GB plus SB will be performed. In case of a Gleason score upgrading by the targeted biopsy the patient will discontinue AS and get treatment. In cases of stable MRI or stable Gleason score the patient will continue with PSA controls every 3 months.

In addition all patients with stable PSA values will undergo a mp-MRI after 12 months. If this MRI demonstrates progression the protocol proceeds as mentioned above for patients with PSA-increase. At the end of study (24 months after enrollment), all patients will receive another mp-MRI and FUS-GB+SB.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Gleason score of 3+3=6 or 3+4=7a and ≤ 33% of positive biopsy cores verified by an at least 12 core systematic prostate biopsy (SB)
* Organ-confined disease (≤cT2a), note: tumor-positive biopsies in both lobes with non-palpable tumor are rated as cT1c
* PSA value ≤10 ng/ml

Exclusion Criteria:

* Gleason score ≥4+3=7b or a Gleason score 3+4=7a with positive biopsy cores >33% of all cores in SB
* PSA >10 ng/ml
* Patients not able to give informed consent
* Contraindication to mp-MRI
* Contraindication to prostate biopsy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of the discontinuation of Active Surveillance (AS) | 24 months
  Reduction of the discontinuation of AS from 25% to 15% of patients after 24 months based on re-biopsy Gleason score upgrading

SECONDARY OUTCOMES:
Value of MRI (ADC) regarding aggressiveness | 36 months
  Evaluation of ADC values in s/mm2
Detectionrates of targeted (FUS-GB) versus systematic (TRUS-GB) biopsies | 36 months
  Comparison of detection rates (in %)
Detectionrates of targeted (FUS-GB) versus systematic (TRUS-GB) biopsies | 36 months
  Comparison of Gleason score upgrades (in %) (Gleason score in units 6-10 )
Correlation of clinical parameters with Gleason score progression or MRI quantified progression | 36 months
  Correlation of PSA elevation in ng/ml
Correlation of clinical parameters with Gleason score progression or MRI quantified progression | 36 months
  Correlation of PSA density in ng/ml/ml
Correlation of clinical parameters with Gleason score progression or MRI quantified progression | 36 months
  Correlation of age in years
Patient compliance to recommended MRI-based observation | 36 months
  Number of patients drop outs
Patient compliance to recommended MRI-based observation | 36 months
  Patient discontinuation rate (in %)
Evaluation of Resolve DWI | 36 months
  Improvement of SNR (signal-to-noise ratio)
Evaluation of Resolve DWI | 36 months
  Subjective Image Quality (5-point scale; evaluated by 2 blinded radiologists; total score from 1=non diagnostic, 2=poor, 3=acceptable, 4=good, to 5=excellent)
Evaluation of Resolve DWI | 36 months
  Improvement of tumor detection rate (in %)
Evaluation of Resolve DWI | 36 months
  NPV (in %)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Schimmöller, MD, Principal Investigator — University Düsseldorf, Medical Faculty; Department of Diagnostic and Interventional Radiology; Christian Arsov, MD, Principal Investigator — University Düsseldorf, Medical Faculty; Department of Urology
Locations (1):
- University Düsseldorf, Medical Faculty, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided